CLINICAL TRIAL: NCT03008200
Title: Fetal Pulmonary Artery Acceleration to Ejection Time Ratio (PATET) in the Prediction of Subsequent Development of Respiratory Distress Syndrome (RDS)
Status: Completed | Type: Observational
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Emre Destegül, Pincipal Investigator, Kayseri Education and Research Hospital
Other Study IDs: KayseriEAH
Record Dates: First submitted 2016-12-20; First posted 2017-01-02 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: RDS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- RDS +: postpartum RDS developed group
  Interventions: Device: ultrasound examination
- RDS -: postpartum RDS undeveloped group
  Interventions: Device: ultrasound examination

INTERVENTIONS:
Device: ultrasound examination — intrauterine fetal pulmonary artery acceleration time to ejection time ratio measurement via ultrasound

SUMMARY:
Fetal PATET ratio evaluation to predict neonatal RDS

DETAILED DESCRIPTION:
115 patients were enrolled in this study.Population was recruited from singleton pregnancies beyond 27 weeks of gestation.All participants underwent a ultrasound examination to measure fetal pulmonary artery acceleration to ejection time ratio (PATET) by a single experienced clinician. After the delivery respiratory distress diagnosis made by a pediatrician who were blinded the doppler waveform measurements.Following the diagnosis, neonates divided into 2 groups as RDS (+) and RDS (-). In addition of RDS diagnosis, neonatal features like 1st and 5th minute APGAR scores, neonatal intensive care unit (NICU) admission and duration in NICU were also recorded. Afterwards all parameters were statistically analyzed if there is any significant differences between those two groups.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women within the 27 weeks of gestation and beyond

Exclusion Criteria:

* patients who did not give birth within 3 days after the ultrasonographic doppler examination
* fetuses with Any congenital abnormalities
* amniotic fluid abnormalities
* any chronic maternal diseases or pregnancy complications such as;gestational diabetes mellitus,preeclampsia

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women beyond 27 weeks
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2015-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Measurement of fetal pulmonary acceleration time to ejection time ratio via ultrasonography in the 115 pregnant women between 27 to 37 weeks of gestation for prediction of respiratory distress syndrome | Ten months
  The aim of this study is to obtain the effectiveness of fetal pulmonary artery acceleration time to ejection time ratio in fetal lung maturity evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Barıs Buke, Principal Investigator — Kayseri Education and Research Hospital

IPD SHARING:
Plan to Share IPD: Yes
if necessary

REFERENCES:
- [Background] Schenone MH, Samson JE, Jenkins L, Suhag A, Mari G. Predicting fetal lung maturity using the fetal pulmonary artery Doppler wave acceleration/ejection time ratio. Fetal Diagn Ther. 2014;36(3):208-14. doi: 10.1159/000358299. Epub 2014 Aug 13. PMID 25139576
- [Background] Azpurua H, Norwitz ER, Campbell KH, Funai EF, Pettker CM, Kleine M, Bahtiyar MO, Malkus H, Copel JA, Thung SF. Acceleration/ejection time ratio in the fetal pulmonary artery predicts fetal lung maturity. Am J Obstet Gynecol. 2010 Jul;203(1):40.e1-8. doi: 10.1016/j.ajog.2010.01.075. Epub 2010 Apr 24. PMID 20417479
- [Background] Guan Y, Li S, Luo G, Wang C, Norwitz ER, Fu Q, Tu X, Tian X, Zhu J. The role of doppler waveforms in the fetal main pulmonary artery in the prediction of neonatal respiratory distress syndrome. J Clin Ultrasound. 2015 Jul-Aug;43(6):375-83. doi: 10.1002/jcu.22219. Epub 2014 Aug 11. PMID 25110859